CLINICAL TRIAL: NCT00547911
Title: L-Dihydroxyphenylserine (L-DOPS) for Norepinephrine Deficiency: Interactions With Carbidopa and Entacapone
Brief Title: Augmenting Effects of L-DOPS With Carbidopa and Entacapone
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study terminated due to contamination droxidopa
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 080012; 08-N-0012 (Other: NIH)
Record Dates: First submitted 2007-10-19; First posted 2007-10-23 (Estimated); Results first posted 2014-07-17 (Estimated); Last update posted 2014-07-17 (Estimated); Status verified 2014-06

CONDITIONS: Parkinson Disease; Multiple System Atrophy; Autonomic Nervous System Diseases
Keywords: Entacapone; Carbidopa; Locus Ceruleus/Norepinephrine-Autonomic System; Norepinephrine; Adrenergic Nervous System
MeSH Terms: conditions — Parkinson Disease; Multiple System Atrophy; Autonomic Nervous System Diseases | interventions — Droxidopa; Carbidopa; entacapone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- LDOPS + Placebo; LDOPS + CAR; LDOPS + ENT (Experimental): Each subject received 400 mg of droxidopa (LDOPS) with three separate interventions, i.e., LDOPS with 200 mg placebo, LDOPS with 200 mg carbidopa (CAR), and LDOPS with 200 mg entacapone (ENT). The order of the three interventions was randomly assigned prior to drug administration and each intervention was followed by a wash out period of at least two days. This arm received the three interventions in the order of: LDOPS + Placebo, followed by LDOPS + CAR, followed by LDOPS + ENT.
  Interventions: Drug: Droxidopa; Drug: Carbidopa; Drug: Entacapone
- LDOPS + Placebo; LDOPS + ENT; LDOPS + CAR (Experimental): There are three interventions that every subject orally received over the duration of the study; 400 mg of droxidopa (LDOPS) + 200 mg placebo, 400 mg of droxidopa (LDOPS) + 200 mg carbidopa (CAR), and 400 mg of droxidopa (LDOPS) + 200 mg entacapone (ENT). The order of the three interventions was randomly assigned prior to drug administration and each intervention was followed by a wash out period of at least two days to clear previous intervention from subject's systems. This arm received the three interventions in the order of: LDOPS + Placebo, followed by LDOPS + ENT, and lastly LDOPS + CAR.
  Interventions: Drug: Droxidopa; Drug: Carbidopa; Drug: Entacapone
- LDOPS + CAR; LDOPS + Placebo; LDOPS + ENT (Experimental): There are three interventions that every subject orally received over the duration of the study; 400 mg of droxidopa (LDOPS) + 200 mg placebo, 400 mg of droxidopa (LDOPS) + 200 mg carbidopa (CAR), and 400 mg of droxidopa (LDOPS) + 200 mg entacapone (ENT). The order of the three interventions was randomly assigned prior to drug administration and each intervention was followed by a wash out period of at least two days to clear previous intervention from subject's systems. This arm received the three interventions in the order of: LDOPS + CAR, followed by LDOPS + Placebo, and lastly LDOPS + ENT.
  Interventions: Drug: Droxidopa; Drug: Carbidopa; Drug: Entacapone
- LDOPS + CAR; LDOPS + ENT; LDOPS + Placebo (Experimental): There are three interventions that every subject orally received over the duration of the study; 400 mg of droxidopa (LDOPS) + 200 mg placebo, 400 mg of droxidopa (LDOPS) + 200 mg carbidopa (CAR), and 400 mg of droxidopa (LDOPS) + 200 mg entacapone (ENT). The order of the three interventions was randomly assigned prior to drug administration and each intervention was followed by a wash out period of at least two days to clear previous intervention from subject's systems. This arm received the three interventions in the order of: LDOPS + CAR, followed by LDOPS + ENT, and lastly LDOPS + Placebo.
  Interventions: Drug: Droxidopa; Drug: Carbidopa; Drug: Entacapone
- LDOPS + ENT; LDOPS + Placebo; LDOPS + CAR (Experimental): There are three interventions that every subject orally received over the duration of the study; 400 mg of droxidopa (LDOPS) + 200 mg placebo, 400 mg of droxidopa (LDOPS) + 200 mg carbidopa (CAR), and 400 mg of droxidopa (LDOPS) + 200 mg entacapone (ENT). The order of the three interventions was randomly assigned prior to drug administration and each intervention was followed by a wash out period of at least two days to clear previous intervention from subject's systems. This arm received the three interventions in the order of: LDOPS + ENT, followed by LDOPS + Placebo, and lastly LDOPS + CAR.
  Interventions: Drug: Droxidopa; Drug: Carbidopa; Drug: Entacapone
- LDOPS + ENT; LDOPS + CAR; LDOPS + Placebo (Experimental): There are three interventions that every subject orally received over the duration of the study; 400 mg of droxidopa (LDOPS) + 200 mg placebo, 400 mg of droxidopa (LDOPS) + 200 mg carbidopa (CAR), and 400 mg of droxidopa (LDOPS) + 200 mg entacapone (ENT). The order of the three interventions was randomly assigned prior to drug administration and each intervention was followed by a wash out period of at least two days to clear previous intervention from subject's systems. This arm received the three interventions in the order of: LDOPS + ENT, followed by LDOPS + CAR, and lastly LDOPS + Placebo.
  Interventions: Drug: Droxidopa; Drug: Carbidopa; Drug: Entacapone

INTERVENTIONS:
Drug: Droxidopa
  Other Names: L-DOPS; Northera; L-threo-dihydroxyphenylserine; SM-5688
Drug: Carbidopa
  Other Names: Lodosyn
Drug: Entacapone
  Other Names: Comtan

SUMMARY:
An experimental drug called L-DOPS increases production in the body of a messenger chemical called norepinephrine. Cells in the brain that make norepinephrine are often gone in Parkinson disease. The exact consequences of this loss are unknown, but they may be related to symptoms such as fatigue, depression, or decreased attention that occur commonly in Parkinson disease. This study will explore effects of L-DOPS in conjunction with carbidopa and entacapone, which are drugs used to treat Parkinson disease. We wish to find out what the effects are of increasing norepinephrine production in the brain and whether carbidopa and entacapone augment those effects.

Volunteers for this study must be at least 18 years of age and able to give consent to participate in the study. To participate in the study, volunteers must discontinue use of alcohol, tobacco, and certain herbal medicines or dietary supplements, and must also taper or discontinue certain kinds of medications that might interfere with the results of the study. Candidates will be screened with a medical history and physical exam.

Participants will be admitted to the National Institutes of Health Clinical Center for two weeks of testing. The study will have three testing phases in a randomly chosen order for each participant:

* Single dose of L-DOPS
* Single dose of L-DOPS in conjunction with carbidopa
* Single dose of L-DOPS in conjunction with entacapone

Each phase will last two days, with a washout day between each phase in which no drugs will be given and no testing will be performed. In each phase, participants will undergo a series of tests and measurements, including blood pressure and electrocardiogram tests. Participants who are healthy volunteers will also have blood drawn and will undergo a lumbar puncture (also known as a spinal tap) to obtain spinal fluid for chemical tests.

DETAILED DESCRIPTION:
Objective: L-DOPS is a synthetic chemical that can be converted to norepinephrine (NE). NE is a key messenger of the sympathetic nervous system. Failure of the sympathetic nervous system results in orthostatic hypotension (OH), a fall in blood pressure when the person stands up. Patients with Parkinson disease (PD) often have OH that is related to loss of sympathetic nerves and to NE deficiency. L-DOPS can help treat OH in these patients. Drugs used commonly to treat PD, however, probably influence effects of L-DOPS. Carbidopa, which combined with levodopa (brand name Sinemet) is a standard treatment for PD, might prevent L-DOPS from being turned into NE outside the brain and therefore interfere with effects of L-DOPS on blood pressure. Entacapone (brand name Comtan) might augment production of NE after a dose of L-DOPS, by decreasing metabolic breakdown of L-DOPS. The first goal of this study is to test these hypotheses in patients with neurogenic OH. NE is also a chemical messenger in the brain and is thought to participate in a variety of neuropsychiatric phenomena such as vigilance, mood, memory, and transmission of pain sensation. Patients with OH can have evidence of central NE deficiency. A second goal of this study is to determine whether depressed mood, apathy, fatigue, or pain improve with L-DOPS treatment in these patients. A third goal is to test whether carbidopa and entacapone, which both should enhance delivery of L-DOPS to the brain, augment L-DOPS effects on these symptoms. Finally, a fourth goal is to verify that carbidopa and entacapone augment neurochemical indices of central neural production of NE after a dose of L-DOPS.

Study Population: The subjects are patients with PD+NOH, MSA+NOH, or pure autonomic failure (PAF); and healthy volunteers. A total of 55 patients and 15 healthy volunteers are to be enrolled.

Design: Patients and healthy volunteers enter this Protocol after undergoing clinical laboratory evaluation under NIH Clinical Protocol 03-N-0004, to confirm the diagnosis, identify NOH, and provide data related to central or peripheral NE production. Each subject serves as his or her own control. Subjects are tested after taking a single oral dose of 400 mg of L-DOPS in a randomized crossover design study of three treatment conditions L-DOPS alone, L-DOPS after carbidopa (200 mg), and L-DOPS after entacapone (200 mg). Healthy volunteers have CSF drawn by lumbar puncture under fluoroscopic guidance about 3 hours after administration of each drug combination.

Outcome Measures:

Primary: Hemodynamics, plasma catechols and their metabolites, non-motor symptom checklists

Secondary: (In healthy volunteers) CSF catechols and their metabolites

Other: (In patients with dysarthria) Speech

ELIGIBILITY:
* INCLUSION CRITERIA:

All subjects in this Protocol will have already undergone clinical laboratory evaluations called for in Clinical Protocol 03-N-0004, "Clinical Laboratory Evaluation of Primary Chronic Autonomic Failure.

EXCLUSION CRITERIA:

Age: People younger than 18 years old are excluded.

Risk: A candidate subject is excluded if, in the judgment of the Principal Investigator or Clinical Director, Protocol participation would place the subject at substantially increased acute medical risk. This includes the risks associated with air travel to the NIH. A candidate subject is excluded if, in the opinion of the Principal Investigator or Clinical Director, the medical risk outweighs the potential scientific benefit.

Disqualifying Conditions: A candidate subject is excluded if there is a disqualifying condition. Examples of disqualifying conditions are hepatic or renal failure, symptomatic congestive heart failure, severe anemia, psychosis, refractory ventricular arrhythmias, and symptomatic coronary heart disease. Persons with dementia interfering with their ability to provide informed consent are excluded. If dementia is suspected, such as by score on the mini-mental examination of less than 24, then a bioethics consult will be obtained.

Medications: A candidate subject is excluded if clinical considerations require that the patient continue treatment with a drug likely to interfere with the scientific results. Examples would be treatment with levodopa/carbidopa or a tricyclic antidepressant. Patients with known or suspected allergy or hypersensitivity to any test drug are excluded. Patients unable to discontinue nicotine or alcohol temporarily are excluded. Patients are not to discontinue any medications before the patient or the patient s doctor discusses this with Dr. Goldstein, the Principal Investigator, or Sandra Pechnik, the Research Nurse. If it is decided that discontinuing medications would be unsafe, then the patient is excluded from the study. Subjects must discontinue use of alcohol and tobacco throughout the period of testing. PD patients who have difficulty tolerating withdrawal of levodopa/carbidopa treatment may be treated with a dopamine receptor agonist during the study, with the dosing remaining the same.

Tricyclic antidepressants, drugs that inhibit L-aromatic-amino-acid decarboxylase or catechol-O-methyltransferase, levodopa, and carbidopa will be withdrawn throughout the period of study. Withdrawal of antiparkinsonian medications may worsen rigidity, bradykinesia, or tremor. These effects are not thought to adversely influence the long-term course of the disease. Withdrawal of tricyclic antidepressants may worsen depression. Drug withdrawal will be done only in inpatients. Alternative drugs, such as serotonin reuptake blockers, anti-anxiety agents, or dopamine receptor agonists, may be used at constant doses during the study.

Herbal Medicines and Dietary Supplements: Certain herbal medicines or dietary supplements are known or suspected to interfere with the experimental results, and such herbal medicines or dietary supplements must be discontinued before enrollment in the study. For many herbal medicines or dietary supplements, the mechanisms of action and therefore the possible effects on the experimental results are unknown. In cases where the subjects wish to continue their herbal medicines or dietary supplements while on study, and search of the available medical literature fails to identify effects that are known or expected to interfere with the experimental results, then the subjects may participate.

Practical Limitations: Subjects in whom we feel it would be difficult to insert a catheter into a vein are excluded. Subjects who are not expected clinically to tolerate lying still supine during the testing are excluded.

Pregnancy: Pregnant or lactating women are excluded. Women of childbearing potential must have a negative urine or blood test for pregnancy done within 24 hours before any testing involving radioactivity or an experimental drug.

Post-Lumbar Puncture Headache: Candidate Healthy Volunteers are excluded if they had a headache requiring a blood patch after lumbar puncture under fluoroscopic guidance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2007-10; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David S Goldstein, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] BLASCHKO H, BURN JH, LANGEMANN H. The formation of noradrenaline from dihydroxyphenylserine. Br J Pharmacol Chemother. 1950 Sep;5(3):431-7. doi: 10.1111/j.1476-5381.1950.tb00593.x. No abstract available. PMID 14777867
- [Background] Halliday GM, Li YW, Blumbergs PC, Joh TH, Cotton RG, Howe PR, Blessing WW, Geffen LB. Neuropathology of immunohistochemically identified brainstem neurons in Parkinson's disease. Ann Neurol. 1990 Apr;27(4):373-85. doi: 10.1002/ana.410270405. PMID 1972319
- [Background] Rajput AH, Rozdilsky B. Dysautonomia in Parkinsonism: a clinicopathological study. J Neurol Neurosurg Psychiatry. 1976 Nov;39(11):1092-100. doi: 10.1136/jnnp.39.11.1092. PMID 188990

RESULTS

PARTICIPANT FLOW:
Groups:
- LDOPS + Placebo; LDOPS + CAR; LDOPS + ENT: There are three interventions that every subject orally received over the duration of the study; 400 mg of droxidopa (LDOPS) + 200 mg placebo, 400 mg of droxidopa (LDOPS) + 200 mg carbidopa (CAR), and 400 mg of droxidopa (LDOPS) + 200 mg entacapone (ENT). The order of the three interventions was randomly assigned prior to drug administration and each intervention was followed by a wash out period of at least two days to clear previous intervention from subject's systems. This arm received the three interventions in the order of: LDOPS + Placebo, followed by LDOPS + CAR, and lastly LDOPS + ENT.
Period: Overall Study
Arm/Group | LDOPS + Placebo; LDOPS + CAR; LDOPS + ENT | LDOPS + Placebo; LDOPS + Ent; LDOPS + CAR | LDOPS + CAR; LDOPS + Placebo; LDOPS + ENT | LDOPS + CAR; LDOPS + ENT; LDOPS + Placebo | LDOPS + ENT; LDOPS + Placebo; LDOPS + CAR | LDOPS + ENT; LDOPS + CAR; LDOPS + Placebo
Started | 2 | 2 | 2 | 2 | 3 | 3
Completed | 2 | 2 | 2 | 1 | 3 | 3
Not Completed | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Healthy Volunteer: Subjects in good general health
- Pure Autonomic Failure: Subjects with Pure Autonomic Failure
- Multiple System Atrophy: Subjects with autonomic failure and a history of Multiple System Atrophy
- Parkinson's Disease: Subjects with autonomic failure and a history of Parkinson's Disease
- Total: Total of all reporting groups
Arm/Group | Healthy Volunteer | Pure Autonomic Failure | Multiple System Atrophy | Parkinson's Disease | Total
Number analyzed (Participants) | 2 | 7 | 2 | 3 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.5 (1.5) | 68.6 (8.1) | 57.0 (0) | 65.0 (7.1) | 64.0 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 1 | 1 | 4
  Male | 2 | 5 | 1 | 2 | 10

OUTCOME MEASURES:

1. Primary Outcome: Plasma LDOPS Concentrations After 400 mg of Droxidopa + 200 mg of Either Placebo, Carbidopa, or Entacapone
Description: Blood samples were obtained at baseline and after drug administration at 1 hour, 2 hours, 3 hours, 6 hours, 24 hours, and 48 hours to assess plasma droxidopa (LDOPS) concentrations.
Time Frame: Up to 48 hours after receiving drug(s)
Population: Data for Healthy Volunteers and all Patient groups was combined for analysis due to the low N-value because of premature study termination, which is further described in the "Limitations and Caveats" section. In addition, some subject data was unable to be analyzed due to unreliable measurements.
Measure: Mean (Standard Error); unit: nmol/L
Groups:
- LDOPS + Placebo: Orally received 400 mg of droxidopa after 200 mg of placebo
- LDOPS + CAR: Orally received 400 mg of droxidopa after 200 mg of carbidopa
- LDOPS + ENT: Orally received 400 mg of droxidopa after 200 mg of entacapone
Arm/Group | LDOPS + Placebo | LDOPS + CAR | LDOPS + ENT
Number analyzed (Participants) | 13 | 13 | 14
nmol/L
  Baseline | 0 (0) | 0.003 (0.003) | 0.897 (0.753)
  1 Hour | 2246 (611) | 1731 (440) | 2068 (413)
  2 Hour | 7067 (1955) | 7077 (1324) | 9114 (1962)
  3 Hour | 8695 (1659) | 9059 (1447) | 12008 (2294)
  6 Hour | 6843 (1080) | 7242 (1749) | 7172 (891)
  24 Hour | 211 (103) | 188 (51) | 331 (203)
  48 Hour | 8 (4) | 7 (2) | 6 (1)

2. Primary Outcome: Plasma Norepinephrine Concentrations After 400 mg of Droxidopa + 200 mg of Either Placebo, Carbidopa, or Entacapone
Description: Blood samples were obtained at baseline and after drug administration at 1 hour, 2 hours, 3 hours, 6 hours, 24 hours, and 48 hours to assess plasma norepinephrine concentrations.
Time Frame: Up to 48 hours after receiving drug(s)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: nmol/L
Groups:
- LDOPS + ENT: Orally received 400 mg of droxidopa after 200 mg of carbidopa
Arm/Group | LDOPS + Placebo | LDOPS + CAR | LDOPS + ENT
Number analyzed (Participants) | 13 | 13 | 14
nmol/L
  Baseline | 0.87 (0.19) | 0.85 (0.15) | 1.08 (0.23)
  1 Hour | 0.89 (0.14) | 0.87 (0.16) | 1.06 (0.16)
  2 Hour | 1.17 (0.15) | 0.98 (0.19) | 1.49 (0.16)
  3 Hour | 1.27 (0.15) | 1.12 (0.19) | 1.69 (0.16)
  6 Hour | 1.26 (0.18) | 0.98 (0.19) | 1.62 (0.13)
  24 Hour | 0.85 (0.16) | 0.89 (0.15) | 1.09 (0.19)
  48 Hour | 0.70 (0.13) | 0.85 (0.16) | 0.84 (0.15)

3. Primary Outcome: Plasma DHMA Concentrations After 400 mg of Droxidopa + 200 mg of Either Placebo, Carbidopa, or Entacapone
Description: Blood samples were obtained at baseline and after drug administration at 1 hour, 2 hours, 3 hours, 6 hours, 24 hours, and 48 hours to assess plasma droxymandelic acid (DHMA) concentrations.
Time Frame: Up to 48 hours after receiving drug(s)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | LDOPS + Placebo | LDOPS + CAR | LDOPS + ENT
Number analyzed (Participants) | 13 | 9 | 11
nmol/L
  Baseline | 0.1 (0.1) | 1.66 (0.48) | 0.97 (0.40)
  1 Hour | 4.0 (1.0) | 2.54 (0.49) | 4.58 (1.37)
  2 Hour | 10.1 (5.7) | 1.52 (0.49) | 15.04 (3.76)
  3 Hour | 11.0 (5.1) | 1.70 (0.28) | 19.91 (4.59)
  6 Hour | 15.7 (4.3) | 1.74 (0.33) | 33.03 (10.91)
  24 Hour | 1.4 (0.8) | 3.24 (0.54) | 2.21 (1.11)
  48 Hour | 0.9 (0.4) | 3.00 (0.58) | 0.90 (0.47)

4. Primary Outcome: Plasma DHPG Concentrations After 400 mg of Droxidopa + 200 mg of Either Placebo, Carbidopa, or Entacapone
Description: Blood samples were obtained at baseline and after drug administration at 1 hour, 2 hours, 3 hours, 6 hours, 24 hours, and 48 hours to assess plasma dihydroxyphenylglycol (DHPG) concentrations.
Time Frame: Up to 48 hours after receiving drug(s)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: nmol/L
Groups:
- LDOPS + CAR: Orally received 400 mg of droxidopa after 200 mg of placebo
Arm/Group | LDOPS + Placebo | LDOPS + CAR | LDOPS + ENT
Number analyzed (Participants) | 13 | 14 | 14
nmol/L
  Baseline | 3.4 (0.4) | 3.4 (0.4) | 3.5 (0.3)
  1 Hour | 4.1 (0.6) | 3.5 (0.4) | 8.0 (1.2)
  2 Hour | 5.4 (0.9) | 3.3 (0.5) | 16.6 (2.3)
  3 Hour | 6.1 (0.8) | 3.6 (0.6) | 19.3 (3.2)
  6 Hour | 5.7 (0.8) | 3.5 (0.8) | 10.7 (1.6)
  24 Hour | 3.4 (0.5) | 3.8 (0.4) | 4.1 (0.4)
  48 Hour | 3.4 (0.4) | 3.7 (0.5) | 3.8 (0.3)

5. Secondary Outcome: Systolic Blood Pressures After 400 mg of Droxidopa + 200 mg of Either Placebo, Carbidopa, or Entacapone
Description: Systolic blood pressure was assessed at baseline and after drug administration at 1 hour, 2 hours, 3 hours, 6 hours, and 24 hours.
Time Frame: Up to 24 hours after receiving drug(s)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | LDOPS + Placebo | LDOPS + CAR | LDOPS + ENT
Number analyzed (Participants) | 13 | 14 | 13
mmHg
  Baseline | 140 (7) | 143 (6) | 139 (5)
  1 Hour | 148 (8) | 144 (7) | 149 (8)
  2 Hour | 163 (10) | 144 (11) | 158 (10)
  3 Hour | 165 (10) | 148 (8) | 161 (12)
  6 Hour | 161 (9) | 146 (8) | 159 (9)
  24 Hour | 149 (7) | 143 (6) | 144 (7)

6. Secondary Outcome: Diastolic Blood Pressures After 400 mg of Droxidopa + 200 mg of Either Placebo, Carbidopa, or Entacapone
Description: Diastolic blood pressure was assessed at baseline and after drug administration at 1 hour, 2 hours, 3 hours, 6 hours, and 24 hours.
Time Frame: Up to 24 hours after receiving drug(s)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | LDOPS + Placebo | LDOPS + CAR | LDOPS + ENT
Number analyzed (Participants) | 13 | 14 | 13
mmHg
  Baseline | 80 (4) | 81 (4) | 78 (4)
  1 Hour | 85 (5) | 80 (5) | 85 (5)
  2 Hour | 86 (6) | 81 (6) | 91 (5)
  3 Hour | 88 (7) | 84 (5) | 91 (6)
  6 Hour | 89 (5) | 82 (5) | 89 (5)
  24 Hour | 84 (3) | 81 (4) | 81 (3)

7. Secondary Outcome: Heart Rate After 400 mg of Droxidopa + 200 mg of Either Placebo, Carbidopa, or Entacapone
Description: Heart rate was assessed at baseline and after drug administration at 1 hour, 2 hours, 3 hours, 6 hours, and 24 hours.
Time Frame: Up to 24 hours after receiving drug(s)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: BPM
Arm/Group | LDOPS + Placebo | LDOPS + CAR | LDOPS + ENT
Number analyzed (Participants) | 13 | 14 | 14
BPM
  Baseline | 67 (3) | 66 (3) | 67 (3)
  1 Hour | 65 (3) | 68 (4) | 65 (2)
  2 Hour | 66 (3) | 65 (3) | 65 (3)
  3 Hour | 68 (4) | 64 (3) | 64 (3)
  6 Hour | 67 (4) | 62 (2) | 67 (2)
  24 Hour | 66 (3) | 66 (3) | 68 (4)

ADVERSE EVENTS:
Time Frame: Duration of the study
Arm/Group | LDOPS + Placebo; LDOPS + CAR; LDOPS + ENT | LDOPS + Placebo; LDOPS + Ent; LDOPS + CAR | LDOPS + CAR; LDOPS + Placebo; LDOPS + ENT | LDOPS + CAR; LDOPS + ENT; LDOPS + Placebo | LDOPS + ENT; LDOPS + Placebo; LDOPS + CAR | LDOPS + ENT; LDOPS + CAR; LDOPS + Placebo
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/2 | 1/2 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/2 | 0/2 | 0/3 | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LDOPS + Placebo; LDOPS + CAR; LDOPS + ENT (N=2) | LDOPS + Placebo; LDOPS + Ent; LDOPS + CAR (N=2) | LDOPS + CAR; LDOPS + Placebo; LDOPS + ENT (N=2) | LDOPS + CAR; LDOPS + ENT; LDOPS + Placebo (N=2) | LDOPS + ENT; LDOPS + Placebo; LDOPS + CAR (N=3) | LDOPS + ENT; LDOPS + CAR; LDOPS + Placebo (N=3)
Deep Vein Thrombosis followed by Pulmonary Embolism (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 — Subject experienced SAE while at home after receiving the LDOPS + CAR and LDOPS + ENT but before receiving the LDOPS + Placebo. Subject was discontinued from protocol and it was determined that the SAE was unlikely due to any study procedures.

LIMITATIONS AND CAVEATS:
Study was prematurely terminated due to a small amount of DOPAL contamination in the droxidopa. Because of the early termination only a small number of subjects were enrolled in each condition. Recently, the FDA has approved droxidopa.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes